CLINICAL TRIAL: NCT00366431
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Oral MOA-728 for the Treatment of Opioid-Induced Bowel Dysfunction in Subjects With Chronic Non-Malignant Pain
Brief Title: Study Evaluating Oral MOA-728 for the Treatment of Opioid-Induced Bowel Dysfunction (OIBD) in Subjects With Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3200A3-200
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Constipation
Keywords: OIBD; OIC; Opioid; Constipation; Laxative
MeSH Terms: conditions — Constipation

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
The primary purpose of the protocol is to evaluate the safety, efficacy, and tolerability of MOA-728 in subjects with Opioid-Induced Bowel Dysfunction (OIBD) with associated chronic non-malignant pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients with opioid-induced bowel dysfunction and chronic non-malignant pain.
* Taking oral, transdermal, intravenous, or subcutaneous opioids.
* Willingness to discontinue all pre-study laxative therapy and utilize only study permitted rescue laxatives.

Exclusion Criteria:

* History of chronic constipation before the initiation of opioid therapy.
* Other GI disorders known to affect bowel transit.
* Women who are pregnant, breast-feeding, or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2006-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The effect of the interventional treatment will be measured by the change from baseline in the number of bowel movements per week during the double-blind treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (56):
- United States (56):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Anaheim, California
  - Bakersfield, California
  - Foothill Ranch, California
  - Garden Grove, California
  - Los Gatos, California
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - Trumbull, Connecticut
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Largo, Florida
  - Miami, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Saint Cloud, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Dawsonville, Georgia
  - Marietta, Georgia
  - Bloomington, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Elkridge, Maryland
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Saginaw, Michigan
  - Traverse City, Michigan
  - Picayune, Mississippi
  - Independence, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Reno, Nevada
  - Haddon Heights, New Jersey
  - Albuquerque, New Mexico
  - Great Neck, New York
  - Lake Success, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Clinton, Oklahoma
  - Chattanooga, Tennessee
  - Beaumont, Texas
  - Colleyville, Texas
  - San Antonio, Texas
  - Alexandria, Virginia
  - Christiansburg, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia